CLINICAL TRIAL: NCT02416674
Title: Vascularized Composite Allotransplantation for Treatment of Abdominal Wall Defects
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Bohdan Pomahac, Director, Plastic Surgery Transplantation, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013P002556
Record Dates: First submitted 2015-04-07; First posted 2015-04-15 (Estimated); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Abdominal Wall Defect
Keywords: abdominal wall; vascularized composite allotransplantation
MeSH Terms: interventions — Vascularized Composite Allotransplantation; Immunosuppressive Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Transplant recipients (Experimental): The intervention is transplantatoin of abdominal wall tissues from an organ donor who is deceased to a recipient with a large abdominal wall defect.
  Interventions: Procedure: abdominal wall transplantation; Drug: Immunosuppressive Agents

INTERVENTIONS:
Procedure: abdominal wall transplantation — transfer of abdominal wall tissues from an organ donor to a pacient with a large abdominal wall defect.
  Other Names: vascularized composite allotransplantation
Drug: Immunosuppressive Agents — Recipients of abdominal wall transplants will need to receive global immunosuppression with tacrolimus, mycophenolate mofetil and prednisone.

SUMMARY:
Abdominal wall transplantation surgery is the transfer of abdominal wall tissues from a deceased human donor to a patient with a large abdominal wall defect. Abdominal wall transplantation is an innovative reconstructive procedure that has the potential to significantly improve the lives of patients with large abdominal wall defects. The purpose of this study is to develop the best practices for abdominal wall transplantation that will improve the outcomes of future abdominal wall transplant recipients.

DETAILED DESCRIPTION:
Abdominal wall transplantation surgery, the transfer of the abdominal wall tissues from a deceased human donor to a patient with a large abdominal wall defect, is an experimental reconstructive procedure that has the potential to significantly improve the lives of patients.

In abdominal wall transplantation, the tissues transplanted include skin, tendons, muscles, ligaments, bones and blood vessels. The transplant team at Brigham and Women's Hospital includes a wide variety of medical and surgical specialties.

The team BWH is actively seeking qualified candidates for the abdominal wall transplantation research study. We will be studying a small group of people to learn more about:

* How to advance the science of abdominal wall transplantation
* How to support and limit transplant rejection issues
* How people do after abdominal wall transplantation We describe abdominal wall transplant surgery as a life-giving procedure because it has the potential to dramatically improve, that is to restore, both a patient's mental and physical health and his/her ability to function and integrate in society. However, as with any other type of organ transplantation, this improvement will require the patient to make a lifetime commitment to taking medications that suppress the body's immune system.

Conventional reconstruction methods are always considered first, but they may provide less than optimal results for certain patients. There are other methods available to reconstruct the abdominal wall. However, they may yield unsatisfactory outcomes in some patients. Abdominal wall transplantation surgery, however, has the potential to deliver these desired functional and aesthetic benefits. Functionally, abdominal wall transplant surgery can provide a patient with a new abdominal wall that, after extensive rehabilitation, will provide mobility and a more natural aesthetic appearance.

From the time we begin our search for a qualified abdominal wall transplant recipient to the continuing care we provide following surgery, a significant amount of time, expertise and attentiveness is contributed toward making the procedure a progressive success. Abdominal wall transplant candidates go through an extensive screening process that is likely to last several months. This screening includes a psychiatric and social support evaluation and a series of imaging tests to help determine a patient's physical and mental readiness for the procedure. If, upon completion of the screening process, it is determined that a patient is a suitable candidate, we will place the patient on a transplant waiting list. We will then begin working with the United Network for Organ Sharing to find a donor who matches the recipient's tissue requirements - for example similar age and correct blood type. This search could take many months, and, if a suitable donor is not found within one year, we will speak with the patient to determine whether he/she is willing to continue waiting.

ELIGIBILITY:
Inclusion Criteria:

* Abdominal wall defects as described above
* Strong motivation to proceed with transplantation
* Accepts dedicating at least 2 years towards extensive post transplant rehabilitation
* Age between 18 and 60 years
* Elapsed injury-to-transplant time of more than 6 months and less than 15 years
* Reports sub-optimal outcome with conventional reconstructive procedures
* Normal liver and kidney function tests:

Exclusion Criteria:

* Record of poor compliance
* Unable to receive adequate follow-up care
* Unable to receive immune suppression either due to geographic or financial limitations
* Unable to follow strict rehabilitation schedule.
* Documented psychological disorder(s) or incomplete psychological clearance
* Impaired renal or hepatic function
* Active cancer with or without metastases
* Severe cardiac/pulmonary dysfunction or other severe irreversible/uncorrectable disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2015-03-01 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
allograft survival | 5 years

SECONDARY OUTCOMES:
immune rejection episodes | 5 years
infections | 5 years
donation of abdominal wall | 5 years
  We will investigate how families of deceased organ donors respond to the request for donation of the abdominal wall tissues

CONTACTS AND LOCATIONS:
Overall Officials: Bohdan Pomahac, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No